CLINICAL TRIAL: NCT04500249
Title: SPI-guided Analgesia in Patients Undergoing Carotid Endarterectomy Under Cervical Plexus Block
Brief Title: SPI-guided Analgesia During CEA Under RA
Acronym: CEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Collaborators: Silesian University of Medicine (Other)
Responsible Party: Principal Investigator, Michał Stasiowski, Principal Investigator, 2Department of Anaesthesiology and Intensive Therapy, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SilesianMUKOAiIT4
Record Dates: First submitted 2019-04-14; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Carotid Artery Stenoses
Keywords: Surgical Pleth Index (SPI); Cervical plexus block; Adequacy of Anaesthesia (AoA; State Entropy; Stroke
MeSH Terms: conditions — Carotid Stenosis; Early-onset ataxia with oculomotor apraxia and hypoalbuminemia; Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: neither participant nor operator is aware of rescue analgesia protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPB (Experimental): cervical plexus block was performed with 0,5% bupivacaine using Moore's technique
  Interventions: Drug: infiltration rescue intraoperative analgesia; Drug: rescue IA; Drug: rescue antyhypertensive medication; Drug: rescue antyemetic medication; Drug: rescue antyhypotensive medication
- CPB with SPI guided analgesia (Experimental): cervical plexus block was performed with 0,5% bupivacaine using Moore's technique alongside with SPI-guided rescue analgesia using 1% lidokaine and intravenous fentanyl
  Interventions: Drug: infiltration rescue intraoperative analgesia; Drug: rescue IA; Drug: rescue antyhypertensive medication; Drug: rescue antyemetic medication; Drug: rescue antyhypotensive medication
- CPB plus SPI guided analgesia plus carotid artery block (Experimental): cervical plexus block was performed with 0,5% bupivacaine using Moore's technique combined ith US-guided carotid artery block alongside with SPI-guided rescue analgesia using 1% lidokaine and intravenous fentanyl
  Interventions: Drug: infiltration rescue intraoperative analgesia; Drug: rescue IA; Drug: rescue antyhypertensive medication; Drug: rescue antyemetic medication; Drug: rescue antyhypotensive medication

INTERVENTIONS:
Drug: infiltration rescue intraoperative analgesia — in the case of intraoperative pain perception, rescue infiltration analgesia using 1 % lidocaine administered by the operator into the operation field.
  Other Names: rescue LA
Drug: rescue IA — in the case of intraoperative pain perception, rescue intravenous analgesia using 50 mcg of fentanyl will be administered by anaesthesiologist
Drug: rescue antyhypertensive medication — in the case of intraoperative hypertension reluctant to rescue analgesia, rescue intravenous antihypertensive medication using 10 mcg of urapidil will be administered by anaesthesiologist
Drug: rescue antyemetic medication — in the case of postoperative nausea and vomitting, rescue intravenous antiemetic medication using 4 mg of ondansetron will be administered by anaesthesiologist
Drug: rescue antyhypotensive medication — in the case of intraoperative hypotension, rescue intravenous antihypotensive medication using 10 mg of ephedrine will be administered by anaesthesiologist
Drug: rescue antyhypotensive medication — in the case of intraoperative bradycardia, rescue intravenous antihypotensive medication using 500 mcg of atropine will be administered by anaesthesiologist

SUMMARY:
The aim of this randomized prospective trial is to assess the utility of Adequacy of Anaesthesia technique (Response Entropy and Surgical Pleth Index) for monitoring pain perception intraoperatively, maintainance of hemodynamic stability during anesthesia and its influence on postoperative outcomes, in patients undergoing carotid endarterectomy under cervical plexus block.

DETAILED DESCRIPTION:
Carotid artery stenosis constitutes a major risk factor for ischemic stroke so carotid endarterectomy is performed to protects patients with severe atherosclerotic carotid artery stenosis against stroke.

Surgical Pleth Index (SPI) is reported to properly reflect nociception-antinociception balance in patients undergoing surgical procedures, where a value of 100 corresponds to a high stress level and a value of 0 to a low stress level; values near 50 or increase in value > delta 10 correspond to the stress level which is known to reflect requirement for rescue analgesia.

A randomized interventional trial to evaluate the effects of SPI-guided rescue analgesia on hemodynamic stability during anesthesia in patients undergoing carotid endarterectomy under cervical plexus block.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of stenosis of carotid artery written consent to participate in the study written consent to undergo carotid endarterectomy under regional anaesthesia of cervical plexus using Moore's technique general heath condition I-III of American Society of Anaesthesiology

Exclusion Criteria:

* necessity of administration of vasoactive drugs influencing SPI monitoring pregnancy
* anatomical malformation that make monitoring using SE sensor impossible
* general atherosclerosis and heart rhythm disturbances impairing SPI monitoring
* chronic medication using opioid drugs leading to resistancy to opioids.
* farmacotherapy with anticoagulants
* allergy to local anaesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
haemodynamic stability | intraoperatively
  variations of haemodynamic parametres will be analysed

SECONDARY OUTCOMES:
pain perception using SPI value variations | intraoperatively
  pain perception using SPI value variations will be analysed

OTHER OUTCOMES:
ischaemic stroke | from beginning of operation till discharge from hospital
  presence of ischaemic stroke will be observed
dysarthria | from beginning of operation till discharge from hospital, approximately 2 - 14 days
  presence of dysarthria will be observed
limb paresis | from beginning of operation till discharge from hospital, approximately 2 - 14 days
  presence of limb paresis will be observed
hoarseness | from beginning of operation till discharge from hospital, approximately 2 - 14 days
  presence of hoarseness will be observed
face semiparesis | from beginning of operation till discharge from hospital, approximately 2 - 14 days
  presence of semiparesis will be observed
postoperative nausea and vomitting | from beginning of operation till discharge from hospital, approximately 2 - 14 days
  presence of postoperative nausea and vomitting will be observed

CONTACTS AND LOCATIONS:
Overall Officials: Michał J Stasiowski, M.D, Principal Investigator — Medical University of Silesia
Locations (1):
- Medical University of Silesia, Sosnowiec, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
publication in AiIT
Supporting Information: ICF
Time Frame: within a year
Access Criteria: on a reasonable request

REFERENCES:
- [Result] Gruenewald M, Herz J, Schoenherr T, Thee C, Steinfath M, Bein B. Measurement of the nociceptive balance by Analgesia Nociception Index and Surgical Pleth Index during sevoflurane-remifentanil anesthesia. Minerva Anestesiol. 2015 May;81(5):480-9. Epub 2014 Jul 17. PMID 25032676
- [Result] Gruenewald M, Ilies C, Herz J, Schoenherr T, Fudickar A, Hocker J, Bein B. Influence of nociceptive stimulation on analgesia nociception index (ANI) during propofol-remifentanil anaesthesia. Br J Anaesth. 2013 Jun;110(6):1024-30. doi: 10.1093/bja/aet019. Epub 2013 Mar 6. PMID 23471754
- [Result] Gruenewald M, Ilies C. Monitoring the nociception-anti-nociception balance. Best Pract Res Clin Anaesthesiol. 2013 Jun;27(2):235-47. doi: 10.1016/j.bpa.2013.06.007. PMID 24012235
- [Result] Gruenewald M, Willms S, Broch O, Kott M, Steinfath M, Bein B. Sufentanil administration guided by surgical pleth index vs standard practice during sevoflurane anaesthesia: a randomized controlled pilot study. Br J Anaesth. 2014 May;112(5):898-905. doi: 10.1093/bja/aet485. Epub 2014 Feb 16. PMID 24535604
- [Result] Won YJ, Lim BG, Lee SH, Park S, Kim H, Lee IO, Kong MH. Comparison of relative oxycodone consumption in surgical pleth index-guided analgesia versus conventional analgesia during sevoflurane anesthesia: A randomized controlled trial. Medicine (Baltimore). 2016 Aug;95(35):e4743. doi: 10.1097/MD.0000000000004743. PMID 27583920
- [Result] Calderon AL, Zetlaoui P, Benatir F, Davidson J, Desebbe O, Rahali N, Truc C, Feugier P, Lermusiaux P, Allaouchiche B, Boselli E. Ultrasound-guided intermediate cervical plexus block for carotid endarterectomy using a new anterior approach: a two-centre prospective observational study. Anaesthesia. 2015 Apr;70(4):445-51. doi: 10.1111/anae.12960. Epub 2014 Dec 1. PMID 25440694
- [Result] Tsujikawa S, Ikeshita K. Low-dose dexmedetomidine provides hemodynamics stabilization during emergence and recovery from general anesthesia in patients undergoing carotid endarterectomy: a randomized double-blind, placebo-controlled trial. J Anesth. 2019 Apr;33(2):266-272. doi: 10.1007/s00540-019-02612-w. Epub 2019 Jan 17. PMID 30656404
- [Result] Zdrehus C. Anaesthesia for carotid endarterectomy - general or loco-regional? Rom J Anaesth Intensive Care. 2015 Apr;22(1):17-24. PMID 28913451
- [Result] Ishiguro T, Yoneyama T, Ishikawa T, Yamaguchi K, Kawashima A, Kawamata T, Okada Y. Perioperative and Long-term Outcomes of Carotid Endarterectomy for Japanese Asymptomatic Cervical Carotid Artery Stenosis: A Single Institution Study. Neurol Med Chir (Tokyo). 2015;55(11):830-7. doi: 10.2176/nmc.oa.2014-0398. Epub 2015 Oct 9. PMID 26458845
- [Result] Lee J, Huh U, Song S, Chung SW, Sung SM, Cho HJ. Regional Anesthesia with Dexmedetomidine Infusion: A Feasible Method for the Awake Test during Carotid Endarterectomy. Ann Vasc Dis. 2016;9(4):295-299. doi: 10.3400/avd.oa.16-00049. Epub 2016 Oct 11. PMID 28018501
- [Result] Scimia P, Giordano C, Basso Ricci E, Petrucci E, Fusco P. The ultrasound-guided C2-C4 compartment block combined to dexmedetomidine sedation: an ideal approach for carotid endarterectomy in awake patients. Minerva Anestesiol. 2018 Oct;84(10):1226-1227. doi: 10.23736/S0375-9393.18.12780-5. Epub 2018 Apr 5. No abstract available. PMID 29624030